CLINICAL TRIAL: NCT04789174
Title: Solriamfetol's Effect on Cognitive Health in Apnea Participants During a Randomized Placebo-controlled Study (SHARP): a 5-Week Double-blind, Placebo-controlled, Randomized, Crossover, Multicenter Study of Solriamfetol in Improving Cognitive Function in Participants With Excessive Daytime Sleepiness Associated With Obstructive Sleep Apnea Plus Impaired Cognitive Function
Brief Title: Solriamfetol's Effect on Cognitive Health in Apnea Participants During a Randomized Placebo-controlled Study
Acronym: SHARP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JZP110-405
Record Dates: First submitted 2021-02-25; First posted 2021-03-09 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Excessive Daytime Sleepiness; Obstructive Sleep Apnea; Impaired Cognitive Function
Keywords: Axsome; SHARP; Solriamfetol; EDS; OSA; Cognition; Cognitive Function; DSST
MeSH Terms: conditions — Disorders of Excessive Somnolence; Sleep Apnea, Obstructive | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Solriamfetol (Active Comparator): Solriamfetol 75 mg/d Solriamfetol 150 mg/d
  Interventions: Drug: Solriamfetol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol — Solriamfetol 75 mg/d Solriamfetol 150 mg/d
  Arms: Solriamfetol
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of study JZP110-405 is to determine whether solriamfetol is effective at improving cognitive function in participants with excessive daytime sleepiness (EDS) associated with obstructive sleep apnea (OSA) plus impaired cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 (or the legal age of consent in the jurisdiction in which the study takes place) and 65 years of age, inclusive.
2. Diagnosis of OSA according to International Classification of Sleep Disorders, Third Edition criteria.
3. Participant report (with clinician concurrence) of at least 1 of the following primary OSA therapy criteria:

   * Consistent number of hours of primary PAP therapy use (with downloadable history) for OSA on at least 5 nights/week for at least 1 month prior to Baseline (with or without prior OSA surgical intervention), OR
   * No current use of PAP therapy for at least 1 month prior to Baseline but a history of at least 1 month of attempting to use PAP as the primary OSA therapy with at least 1 documented adjustment that was made in an attempt to optimize the therapy (with or without prior OSA surgical intervention), OR
   * History of a surgical intervention intended to treat OSA symptoms (with or without current PAP use as primary OSA therapy).
4. Usual nightly total sleep time of ≥ 6 hours.
5. Body mass index from 18.5 to < 40 kg/m2.
6. Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 14 days after the last dose of study intervention:

   • Refrain from donating sperm

   PLUS, either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR
   * Must agree to use contraception/barrier
7. A female participant is eligible to participate if she is not pregnant or breastfeeding, and 1 of the following conditions applies:

   * Is a woman of nonchildbearing potential (WONCBP) OR
   * Is a WOCBP and using a contraceptive method that is highly effective
8. Capable of giving signed informed consent.

Exclusion Criteria:

1. Female participants who are pregnant, nursing, or lactating.
2. Usual bedtime later than 1 AM (0100 hours).
3. Occupation requiring nighttime or variable shift work.
4. Unable to understand or perform DSST test per investigator's judgement.
5. Use a PAP machine with no adherence data downloadable ability.
6. Diagnosis of another sleep disorder (other than OSA) including: circadian rhythm sleep disorders, narcolepsy, restless legs syndrome determined by participant sleep history.
7. Presence of acutely unstable major depression or current major depressive episode as based on the judgement of the investigator.
8. Participants with active clinically significant illness, including endocrine, neoplastic, gastrointestinal, hematological, hepatic, immunologic, metabolic, neurological, pulmonary, and/or renal disease, and/or surgical history which could interfere with the study efficacy, safety, conduct or the ability of the participant to complete the study based on the judgement of the investigator, or place the participant at risk during the trial or compromise the study objectives.
9. History or presence of any other clinically relevant medical, behavioral, or psychiatric disorder other than OSA that is associated with an impact on cognitive function.
10. History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
11. History of bariatric surgery within the past year or a history of any gastric bypass procedure.
12. Participants with movement or motor disorders such as Parkinson's disease, as they will not be able to complete the DSST.
13. Presence of renal impairment or calculated creatinine clearance < 60 mL/minute.
14. Clinically significant ECG abnormality in the opinion of the investigator.
15. Presence of significant cardiovascular disease.
16. Laboratory value(s) outside the laboratory reference range that is considered to be clinically significant by the investigator (clinical chemistry, hematology, and urinalysis). NOTE: Screening labs may be repeated once.
17. Hypothyroidism or hyperthyroidism, unless stabilized by appropriate medication for at least 3 months prior to Screening (a normal thyroid-stimulating hormone is required prior to Randomization at Baseline).
18. Use of any over-the-counter (OTC) or prescription medications that could affect the evaluation of EDS within a time period prior to the Baseline visit corresponding to at least 5 half-lives of the drug(s) or planned use of such drug(s) at some point throughout the duration of the 5-week double-blind treatment period.
19. Current or recent (within the past 2 years) diagnosis of a moderate or severe substance use disorder (excluding caffeine) according to DSM-5 criteria, or seeking treatment for a substance-related disorder. Nicotine use disorder is excluded only if it has an effect on sleep (ie, a participant who routinely awakens at night to smoke).
20. Excessive caffeine use.
21. Urine drug screen positive for amphetamine, methamphetamine, tricyclic antidepressants, propoxyphene, benzodiazepines, barbiturates, cocaine, marijuana, morphine, ecstasy, oxycodone, buprenorphine, methadone, or phencyclidine at Screening or at any point throughout the duration of the study.
22. History of regular heavy use of tetrahydrocannabinol (THC) is excluded. Sporadic recreational users of THC can complete a repeat urine drug screen during the Screening period. If this is negative, the participant may be allowed to enter the study pending agreement to completely refrain from the use of THC during the course of the study.
23. Positive alcohol test at Screening.
24. Participants who binge drink, defined as 5 or more drinks in a day for men or 4 or more drinks in a day for women at least once in past month.
25. History of phenylketonuria or history of hypersensitivity to phenylalanine-derived products.
26. Currently receiving MAO inhibitors or having had received MAO inhibitors for 14 days prior to the Baseline visit.
27. Previous exposure to solriamfetol.
28. Received an investigational drug in the past 30 days or 5 half-lives (whichever is longer) prior to the Baseline visit, or plans to use an investigational drug (other than the study drug) during the study.
29. Is currently participating in another clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (15):
  - Southern California Institute for Respiratory Disease, Los Angeles, California
  - SDS Clinical Trials, Inc, Santa Ana, California
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - The Neurological Center of north Georgia., Gainesville, Georgia
  - The Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - Henry Ford Health System, Novi, Michigan
  - Sleep Medicine & Research Center, Chesterfield, Missouri
  - Advanced Respiratory and Sleep Medicine, PLLC, Huntersville, North Carolina
  - CTI-Clinical Research Center, Cincinnati, Ohio
  - Intrepid Research, LLC, Cincinnati, Ohio
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - FutureSearch Trials of Neuroglogy, Austin, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - Sleep and Performance Research Center, Spokane, Washington
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - MedSleep Inc. o/a Toronto Sleep Institute, Toronto, Ontario
  - Jodha Tishon Inc, Toronto, Ontario
- Italy (4):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, Emilia-Romagna
  - IRCCS Ospedale San Raffaele - Servizio Farmacia, Milan, Lombardy
  - IRCCS Associazione Oasi Maria SS Onlus, Troina, Sicily
  - UOC Farmacia e Politiche del farmaco, edif 41, Pisa
- Netherlands (2):
  - Amphia Hospital, Breda
  - Sleep-Waakcentrum SEIN, Heemstede
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Instiut de Reccerca Biomedica de Lledia, Lleida
- Royal Papworh Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Van Dongen HPA, Leary EB, Drake C, Bogan R, Jaeger J, Rosenberg R, Streicher C, Tabuteau H. Results of the Solriamfetol's Effect on Cognitive Health in Apnea Participants During a Randomized Placebo-Controlled Study (SHARP): A Randomized Placebo-Controlled Double-Blind Repeated-Measures Crossover Phase IV Clinical Trial of the Effect of the Wake-Promoting Agent Solriamfetol on Cognitive Function in OSA With Excessive Daytime Sleepiness and Cognitive Impairment. Chest. 2025 Mar;167(3):863-875. doi: 10.1016/j.chest.2024.10.050. Epub 2024 Nov 9. PMID 39528111
- See also: Axsome Therapeutics Website — http://www.axsome.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Crossover Design: Subjects meeting the entry criteria were randomized in a 1:1 ratio either to Sequence 1 (up to 150 mg solriamfetol daily for two weeks followed by placebo for two weeks) or Sequence 2 (placebo for two weeks followed by up to 150 mg solriamfetol daily for two weeks). Crossover treatment periods were separated by a 1-week washout period.
Groups:
- Sequence 1: Sequence 1 - Solriamfetol for two weeks followed by placebo for two weeks
- Sequence 2: Sequence 2 - Placebo for two weeks followed by solriamfetol for two weeks
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2
Started (Started (Safety Population) includes all subjects who received at least one dose of study drug.) | 30 | 29
Dosed With Solriamfetol | 30 | 29
Dosed With Placebo | 30 | 29
mITT Population (mITT Population includes all subjects who received at least one dose of study drug and have at least 1 postdose evaluation of the DSST RBANS.) | 29 | 29
Completed | 29 | 28
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population includes all subjects who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (10.48) | 51.9 (11.10) | 52.2 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 20 | 18 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 24 | 19 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average of the DSST RBANS Scores at the End of Each Double-blind Treatment Period
Description: The DSST RBANS (Digit Symbol Substitution Test Repeatable Battery for the Assessment of Neuropsychological Status) is an objective neuropsychological test that assesses executive function, processing speed and attention. DSST RBANS scores range from a minimum of 0 (worse outcome) to a maximum of 100 (better outcome).
  The change from baseline was calculated as post-baseline - baseline. A positive change indicates improvement.
Time Frame: Baseline to the end of the second double-blind treatment period (up to 5 weeks)
Population: mITT Population includes all subjects who received at least one dose of study drug and have at least 1 postdose evaluation of the DSST RBANS.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Solriamfetol: Solriamfetol dosed daily for up to 2 weeks
- Placebo: Placebo dosed daily for up to 2 weeks
Arm/Group | Solriamfetol | Placebo
Number analyzed (Participants) | 58 | 58
score on a scale | 6.49 (0.650) | 4.75 (0.646)
Statistical Analysis 1: Comparison: Solriamfetol vs Placebo; Test type: Superiority; p = 0.009, Mixed Models Analysis — P-value calculated from LSMean

ADVERSE EVENTS:
Time Frame: Adverse events were collected after administration of study drug through the final visit (up to 6 weeks).
Description: Safety Population includes all subjects who received at least one dose of study drug.
Groups:
- Solriamfetol: Adverse events collected while subjects were in the solriamfetol period of either Sequence 1 or Sequence 2.
- Placebo: Adverse events collected while subjects were in the placebo period of either Sequence 1 or Sequence 2.
Arm/Group | Solriamfetol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 6/59 | 1/59
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solriamfetol (N=59) | Placebo (N=59)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT04789174/Prot_001.pdf
  • Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT04789174/SAP_003.pdf